CLINICAL TRIAL: NCT05756751
Title: IMpella®-Protected cArdiaC Surgery Trial in Europe: A European, Prospective, Multicenter, Post-Market Clinical Follow-Up Trial
Brief Title: IMPACT EU Post-Market Clinical Follow-Up Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABMD-CIP-22-03
Record Dates: First submitted 2023-01-20; First posted 2023-03-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Left Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: Impella 5.5® with SmartAssist® (Impella 5.5®)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment with Impella 5.5 System (Other)
  Interventions: Device: Device: Impella 5.5 with SmartAssist

INTERVENTIONS:
Device: Device: Impella 5.5 with SmartAssist — Patients who are deemed high-risk due to low preoperative ejection fraction undergoing cardiac surgery with cardiopulmonary bypass (CPB) which will be supported by the Impella 5.5 System.

SUMMARY:
The purpose of this trial is to collect further data on the safety and on the effectiveness of the use of Impella 5.5® in high-risk cardiac surgery patients.

DETAILED DESCRIPTION:
A European, prospective, multicenter, post-market clinical single-arm follow-up trial.

Up to 123 patients will be enrolled in the study.

Patients will be followed for up to 1-year.

The objectives of the study are to collect data on the safety and on the effectiveness of the Impella 5.5 System in mitigating post-cardiotomy cardiac failure, as well as improving functional status and quality of life (QoL) in high-risk cardiac surgery patients with severe LV dysfunction in a post-market setting.

ELIGIBILITY:
Inclusion Criteria:

1. Hemodynamically stable patients undergoing one (1) of the following cardiac surgery procedures on CPB including aortic cross-clamping and cardioplegic arrest

   * Isolated CABG
   * Isolated mitral valve repair or replacement (MVR)
   * Isolated aortic valve repair or replacement (AVR)
   * At lest two of the following: CABG, MVR, AVR, or tricuspid valve repair or replacement (TVR)
2. LVEF within 30 days before surgery of either:

   * ≤25% measured by echocardiogram or
   * LVEF ≤35% as above for patients with significant mitral regurgitation (MR 3+ or 4+; see definition) and planned corrective mitral valve surgery (including MV replacement or repair)
3. Age 18 years or older
4. Subject has signed informed consent form and is willing and able to attend all follow-up visits and to perform all tests.
5. Patient is eligible to receive the Impella 5.5 as per the current IFU.

Exclusion Criteria:

1. Salvage operation (cardiac arrest within 24 hours prior to index surgery)
2. Unresponsive state within 24 hours of the time of surgery
3. Any inotrope within 72 hours of surgery
4. Any mechanical MCS device (such as IABP, ECMO, Impella®, CentriMag™ or TandemHeart®) in place prior to informed consent
5. RV dysfunction requiring mechanical or inotropic support preoperatively and/or likely to be needed postoperatively
6. Index procedures requiring total circulatory arrest (TCA), such as aortic arch replacement, planned durable LVAD, durable RVAD, planned right-sided temporary mechanical support of any kind, total artificial heart (TAH), cardiac transplantation, pericardiectomy, pulmonary thromboendarterectomy and septal myectomy
7. Restrictive or obstructive cardiomyopathy, constrictive pericarditis, restrictive pericarditis, pericardial tamponade or other conditions in which cardiac output is dependent on venous return
8. Ventricular septal defect (VSD)
9. Stroke within 30 days of the index cardiac surgical procedure
10. Prior mantle field chest irradiation
11. Prior solid organ or hematologic transplantation (heart, kidney, liver, lung, pancreas, bone marrow) or durable LVAD
12. History of chronic dialysis
13. Pre-existing liver dysfunction defined as Child-Pugh Class B or C
14. Pre-existing pulmonary disease requiring home oxygen, or "severe pulmonary disease" determined by enrolling investigator
15. Systemic active infection or evidence of systemic bacterial, fungal or viral infection within 72 hours before surgery (blood culture positive with leukocytosis)
16. Confirmed COVID-19 infection within two (2) weeks prior to operation
17. Pregnant or planning pregnancy within next 12 months. NOTE: Female patients of childbearing potential need to have a negative pregnancy test performed within 14 days prior to intervention.
18. Participation in the active treatment or follow-up phase of another interventional clinical trial of an investigational drug or device which has not reached its primary endpoint
19. Known contraindication to heparin; History of bleeding diathesis or known coagulopathy or will refuse blood transfusions
20. Inability to perform aortic cross-clamp, such as due to porcelain aorta
21. Any contraindication or condition that would prevent the ability to place Impella 5.5® (per current IFU), including LV thrombus and/or presence of a mechanical aortic valve
22. Any organ condition, concomitant disease (e.g., psychiatric illness, current severe alcoholism or current drug abuse, cancer, hepatic or kidney disease), with life expectancy of ≤2 years or other abnormality that itself or the treatment of which, could interfere with the conduct of the trial or that, in the opinion of the investigator would pose an unacceptable risk to the subject in the trial.
23. Subject has other medical, social or psychological problems that, in the opinion of the investigator, compromises the subject's ability to give written informed consent and/or to comply with trial procedures, including patients under guardianship
24. Any subject considered to be part of a vulnerable population (as per ISO 14155)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
the rate of post-cardiotomy cardiac failure | Through Hospital Discharge, on average 1 week
All-cause mortality | 90 Days after procedure
Stroke (as defined by STS) | 90 Days after procedure
  Postoperative stroke (cerebrovascular accident) consisting of any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain that did not resolve within 24 hours.

SECONDARY OUTCOMES:
New requirement for renal replacement therapy (RRT) | through study completion, an average of 1 year
Number of attempts to wean from CPB | Until CPB was removed, on average 72 hours
Duration of mechanical ventilation | Through ICU Discharge, on average 3 days
Acute Kidney Injury (a modified KDIGO stages 2-3) | Within 7 days or at ICU discharge whichever comes first
Adequate hemodynamic support | Until Pulmonary Artery Catheter was removed, on average 3 days
Vasoactive-inotropic score (VIS) | Through ICU Discharge, on average 3 days
Cardiovascular mortality | Through Hospital Discharge, on average 1 week
Major Hemolysis (defined by MCS-ARC) | Through Hospital Discharge, on average 1 week
Major Vascular Complications (defined by MCS-ARC) | Through Hospital Discharge, on average 1 week
Major Bleeding defined by STS | Through Hospital Discharge, on average 1 week
  Bleeding requiring surgical intervention or fatal bleeding
All-cause Mortality | Up to 1-year post-op

OTHER OUTCOMES:
Technical Success | Time of CPB removed, on average at 72 hours
  The successful use of the Impella 5.5 device will be assessed by the proportion of patients who undergo successful Impella insertion, as well as the proportion of patients demonstrating successful wean off CPB
Length of ICU stay in days | Through ICU discharge, on average 3 days
Length of hospital stay in days | Through Hospital Discharge, on average 1 week
Quality of Life Assessment by Kansas City Cardiomyopathy Questionnaire KCCQ) | 90 days and 1-year post-op
  KCCQ scores are scaled from 0 to 100. Lower scores representing the worse symptoms
Quality of Life by Assessment of physical activity | 90 days and 1-year post-op
  (Katz Activities of Daily Living (ADL). A The summary score ranges from 0 (low function, dependent) to 8 (high function, independent).
Quality of Life (QoL) by assessing the ability to perform tasks necessary to live independently | 90 days and 1-year post-op
  Assessed by LAWTON - BRODY instrumental activities of daily living scale (I.A.D.L.). A summary score ranges from 0 (Low, patient very dependent ) to 6 (high, patient independent)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann Reichenspurner, Prof. Dr. Dr., Principal Investigator — UKE Hamburg; Payam Akhyari, Prof. Dr., Principal Investigator — Westdeutsches Herz- und Gefäßzentrum Essen
Locations (13):
- IKEM Prague, Prague, Czechia
- Germany (12):
  - Universitätsklinikum Heidelberg - Klinik für Herzchirurgie, Heidelberg, Baden-Wurttemberg
  - RWTH Uniklinik Aachen - Klinik für Herzchirurgie, Aachen, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Klinik für Herzchirurgie, Düsseldorf, North Rhine-Westphalia
  - Universitätsmedizin Essen, Westdeutsches Herzzentrum, Klinik für Thorax- und Kardiovaskuläre Medizin, Essen, North Rhine-Westphalia
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Herz- und Gefäßchirurgie, Mainz, RLP
  - Universitätsmedizin Halle/Saale - Klinik für Herzchirurgie, Halle, SA
  - UKSH Campus Kiel - Klinik für Herz- und Gefäßchirurgie, Kiel, Schleswig-Holstein
  - Deutsches Herzzentrum der Charité, Berlin
  - Universitätsklinikum Giessen, Giessen
  - Universitäres Herz- und Gefäßzentrum Hamburg - Klinik und Poliklinik für Herz- und Gefäßchirurgie, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Krankenhaus der Barmherzigen Brüder Trier, Trier